CLINICAL TRIAL: NCT03684824
Title: Accuracy of Ultrasound Markers Versus Biochemical Markers in Prediction of Ovarian Response in Obese Women Undergoing IVF/ICSI Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Maged, professor, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 39
Record Dates: First submitted 2018-09-19; First posted 2018-09-26 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: Invitro Fertilization
MeSH Terms: interventions — Triptorelin Pamoate; Adenosine Monophosphate; Gonadotropins; hMG-IBSA

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- obese group (Other): 100 obese patients with BMI between 30 and 35 who are undergoing IVF/ICSI treatment for infertility
  Interventions: Drug: Long luteal phase GnRH agonist protocol; Drug: Gonadotropins

INTERVENTIONS:
Drug: Long luteal phase GnRH agonist protocol — Pituitary suppression will be done using daily subcutaneous injection of triptorelin acetate ( Decapeptyl 0.1mg, Ferring, Germany). Starting from day 21 of the previous cycle
  Other Names: Decapeptyl 0.1mg amp
Drug: Gonadotropins — Controlled ovarian hyperstimulation will be done using daily intramuscular injection of highly purified Human Menopausal Gonadotrophins (Merional 75 IU/ml, IBSA, Switzerland), starting from day 2-3 of the stimulated cycle, total dose will be adjusted according to patient response
  Other Names: Merional 75 IU/ml, IBSA, Switzerland

SUMMARY:
After detailed history and examination, long luteal protocol will be used for controlled ovarian hyperstimulation, so the patient will start treatment in day 21 of previous cycle, then in the early follicular phase of next cycle day 2-3 will have transvaginal sonography for assessment of total ovarian volume and number of antral follicles measuring (2-10mm) in diameter. On the same day a venous sample will be obtained for the measurement of AMH, basal FSH and E2 levels

DETAILED DESCRIPTION:
After detailed history and examination,A transvaginal ultrasound will be done using a transvaginal transducer with 7.5 MHz.

Each ovary will be measured in 3 planes maximal longitudinal, antero-posterior and transverse diameters, D1, D2 and D3 respectively. And ovarian volume will be calculated using the ellipsoid formula:

V = D1× D2 × D3 × 0.523 The volume of both ovaries will be added for the total basal ovarian volume (BOV).

The mean diameter of the antral follicles will be used by measuring the diameter of the follicle in two perpendicular directions.

The total AFC is calculated by counting the follicles with mean diameter 2-10mm in both ovaries.

• Ovulation induction protocol:- Long luteal phase agonist protocol will be used in all patients. Pituitary suppression will be done using daily subcutaneous injection of triptorelin acetate ( Decapeptyl 0.1mg, Ferring, Germany). Starting from day 21 of the previous cycle.

Controlled ovarian hyperstimulation will be done using daily intramuscular injection of highly purified Human Menopausal Gonadotrophins (Merional 75 IU/ml, IBSA, Switzerland), starting from day 2-3 of the stimulated cycle, total dose will be adjusted according to patient response.

Induction of oocyte maturation will be done using human chorionic gonadotrophins as an intramuscular injection of 10000 IU hCG (Choriomon 5000 i.u, IBSA, Switzerland). When there was sufficient ovarian response that defined as the presence of three or more ovarian follicles with mean diameter 18mm or more. [15]

• Monitoring of the cycle: The response to ovarian stimulation will be monitored by serial transvaginal ultrasound starting on day 6 of stimulation and onwards assessing the ovarian follicles number and diameter, as well as serum E2 level as indicated.

• Oocyte Retriveal: Oocyte retrieval will done (34-36 hours) after hCG injection, by transvaginal guided vacuumed oocyte aspiration using double lumen oocyte aspiration needle for flushing of the follicles.

• Measurement of FSH and E2 Levels: A blood sample will be withdrawn on day (2 - 3) of the menstrual cycle in which the patient will undergo stimulation, for estimation the basal FSH (mIU/ml) , E2 (pg/ml) and AMH (ng/ml) levels.

Both FSH and E2 will be tested using VIDAS equipment, both the FSH and E2 were measured by automated quantitative testing, using the ELFA technique (Enzyme Linked Fluorescent Assay). In the same way, AMH will be tested by Beckman Coulter, using GenII ELISA, USA.

ELIGIBILITY:
Inclusion Criteria:

* Women between 20 and 35 age.
* BMI: 30 -35

Exclusion Criteria:

* Women less than 19 years or more than 35 years.
* BMI less than 30 or more than 35
* Women with Hypothyroidism.
* Women receiving any treatment may reduce their fertility e.g: chemotherapy.
* Women with recurrent IVF failure

Ages: 19 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
number of retrieved oocytes | 34 hours after HCG triggering of ovulation
  number of oocytes retrieved at day of ovum pick up

SECONDARY OUTCOMES:
Clinical pregnancy rate | 14 days after embryo transfer
  Ultrasound detection of intrauterine gestational sac

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed maged, Principal Investigator — Professor
Locations (1):
- Ameer Elsherief, Minya, Egypt